CLINICAL TRIAL: NCT01441726
Title: Palliative and End-of-life Care in Advanced Dementia: Evaluation of a Program of Organization of Care in Long-term Care Settings
Brief Title: Palliative and End-of-life Care in Advanced Dementia: Evaluation of a Program of Organization of Care in Long-term Care
Status: Completed | Type: Observational
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, René Verreault, Professeur titulaire, Laval University
Other Study IDs: MOP-114881
Record Dates: First submitted 2011-09-07; First posted 2011-09-28 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Dementia
Keywords: Advanced dementia; Quality; Terminal care
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Training of staff
- No training of staff

SUMMARY:
Rationale: In Canada, as in most industrialized countries, Alzheimer's disease and other related dementia are increasingly prevalent in older people. At an advanced stage, institutionalization in a long-term care (LTC) setting will be the fate of a majority of patients. A structured palliative care approach is increasingly used for cancer patients, but is still rarely accessible in LTC institutions for older people with advanced or terminal dementia. This approach should include a more systematic detection and treatment of pain and other physical and psychological symptoms during the last weeks of life, as well as better communications between patients, families and care staff, particularly relating to advanced care directives. Objectives: The general objective of this study is to implement and evaluate a multidisciplinary and multidimensional program of palliative and end-of-life care for older persons with terminal dementia in LTC facilities. Methodology: The intervention program will include five components:

1. daily involvement of a nurse from the regular staff in the LTC facility as a change agent;
2. awareness sessions with administrators and staff on the importance of high quality palliative care in dementia;
3. a training program for physicians and all the staff involved in direct care of patients;
4. systematic discussions with families and distribution to families of a document on different aspects of palliative care in dementia;
5. systematic clinical care by regular staff for the control of pain, respiratory symptoms and mouth care. The program will be implemented in two LTC settings (one in Quebec City and one in Sherbrooke, Quebec, Canada), and results will be compared with the LTC control settings where usual care will be applied without implementation of the program.

ELIGIBILITY:
Inclusion Criteria:

Residents with advanced dementia with a score of 7 on the Reisberg scale

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Residents in long term care settings
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2012-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Family satisfaction with terminal care | 1 year
  Family Perception of Care Scale (FPCS): 25-item validated instrument including 4 components, yielding a score from 25 (negative perception) to 175 (highest positive perception of quality of palliative care)
Comfort scale in last two weeks of life | 2 weeks
  Comfort Assessment in Dying with Dementia (CAD-EOL): 14-item validated instrument including 4 sub-scales, yielding a score from 14 (low comfort level) to 42 (highest comfort level).

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de santé et de services sociaux de la Vieille Capitale, Québec, Quebec, Canada